CLINICAL TRIAL: NCT04023487
Title: Evaluation of a Complex Intervention for Young Adults With Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) Study
Brief Title: Evaluation of an Intervention for Young Adults With Diabetes: Resilient, Empowered, Active Living-Telehealth (REAL-T)
Acronym: REAL-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Beth Pyatak, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DK116719 (NIH); 1R01DK116719 (NIH)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1, randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): Resilient, Empowered, Active Living-Telehealth (REAL-T)
  Interventions: Behavioral: Resilient, Empowered, Active Living-Telehealth (REAL-T)
- Usual Care (No Intervention): Participants will continue to have access to routine diabetes care from the provider of their choosing; they will not receive any study-related intervention.

INTERVENTIONS:
Behavioral: Resilient, Empowered, Active Living-Telehealth (REAL-T) — REAL-T is an individually-tailored occupational therapy intervention that focuses on incorporating diabetes self-care into participants' daily habits and routines. Participants receive approximately 12 hours of intervention, delivered via telehealth over 6 months by a licensed occupational therapist with training in diabetes education, motivational interviewing, and the REAL Diabetes intervention protocol.
  Arms: Lifestyle Intervention

SUMMARY:
This study will evaluate (1) the efficacy of REAL-T, a lifestyle-based telehealth intervention, in improving glycemic control (HbA1c) and psychosocial outcomes, (2) which effects are retained over a 6-month follow-up period, and (3) the mediating mechanisms responsible for the intervention's effects. Half of participants will receive REAL-T, while the other half will receive their usual care.

DETAILED DESCRIPTION:
Evaluation of a Complex Behavioral Intervention for Young Adults with Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) Study will address the unmet self-management and psychosocial needs of young adults (YAs) with type 1 diabetes (T1D).

We will conduct a large-scale randomized controlled trial (n=210) to compare the 6-month REAL-T intervention to usual care in improving glycemic control (A1c and continuous glucose monitor-derived measures), psychosocial well-being, and hypothesized intervention mediators. In addition, we will perform health economic analyses to determine the extent to which REAL-T is cost-effective or produces cost savings.

The study's specific aims are as follows:

Aim 1: Evaluate the efficacy of REAL-T in improving glycemic control and psychosocial well-being.

* Hypothesis 1: Over a 6-month intervention period (including 3 and 6 month measures), YAs with T1D who receive REAL-T demonstrate improvements in glycemic control, in comparison to YAs with T1D who receive usual care.
* Hypothesis 2: Over a 6-month period (including 3 and 6 month measures), YAs with T1D who receive REAL-T demonstrate gains in psychosocial well-being in comparison to YAs with T1D who receive usual care.

Aim 2: Assess the post-intervention durability (at 3 and 6 months post-intervention) of REAL-T's effects on glycemic control and psychosocial well-being.

* Hypothesis 1: Among YAs with T1D, improvements in glycemic control that result from REAL-T relative to usual care are maintained at 3 and 6 months post-treatment.
* Hypothesis 2: Among YAs with T1D, improvements in psychosocial well-being that result from REAL-T relative to usual care are maintained at 3 and 6 months post-treatment.

Aim 3: Examine mediating mechanisms of the REAL-T intervention's effects on glycemic control and psychosocial well-being through structural equation modeling (SEM).

* Hypothesis 1: Improvements in diabetes self-care behaviors mediate positive intervention effects on glycemic control and psychosocial well-being.
* Hypothesis 2: Improvements in self-efficacy mediate positive intervention effects on psychosocial well-being and partially mediate positive effects on diabetes self-care behaviors.
* Hypothesis 3: Improvements in habit strength for diabetes self-care behaviors partially mediate positive intervention effects on the performance of diabetes self-care behaviors.

ELIGIBILITY:
Inclusion Criteria:

* T1D for ≥12 months
* A1c ≥7.5% at time of study enrollment
* Age 18-30 yrs. at time of study enrollment
* English or Spanish speaking
* Resides in a state where OT clinicians are licensed, in an area where the participant has access to a local healthcare provider in the event of emergency and can complete data collection in person (when permitted) or via mailings (when required during period of social distance or due to distance from study site)
* Participant has access to a laptop or desktop computer, either their own or loaned by the study (if geographically feasible and permitted given COVID-19 social distancing distractions)
* Willing to participate in 6-month intervention

Exclusion Criteria:

* Currently pregnant or planning to become pregnant within the next 12 months
* Previously received REAL intervention
* Cognitive impairment or severe disability limiting life expectancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pyatak, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- USC Center for Health Professionals, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle Intervention | Usual Care
Started | 104 | 105
Completed | 86 | 90
Not Completed | 18 | 15
Not completed — Lost to Follow-up | 5 | 4
Not completed — Pregnancy | 1 | 2
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Partially completed testing | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Intervention | Usual Care | Total
Number analyzed (Participants) | 104 | 105 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.88 (3.78) | 24.77 (3.62) | 24.33 (3.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 36 | 39 | 75
  Female | 62 | 63 | 125
  Other | 5 | 3 | 8
  Decline to Answer | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latinx | 49 | 42 | 91
  White | 46 | 47 | 93
  Black | 1 | 7 | 8
  Asian | 2 | 2 | 4
  Other | 0 | 4 | 4
  >1 Race/ethnicity | 5 | 3 | 8
  Decline to Answer | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 104 | 105 | 209
Recruitment Source [Count of Participants; unit: Participants]
  Clinic | 40 | 42 | 82
  Social Media (California) | 40 | 40 | 80
  Social Media (Texas) | 14 | 16 | 30
  Social Media (Oregon, Washington, Colorado) | 10 | 7 | 17
Household composition (non-exclusive) [Count of Participants; unit: Participants] — Household Composition (non-exclusive). Participants can be counted more than once in the appropriate category.
  Participants
    Alone | 1 | 4 | 5
    With parents | 50 | 44 | 94
    With roommates | 21 | 22 | 43
    With partner | 39 | 34 | 73
    Missing/Declined to State | 0 | 1 | 1
Household size [Mean (Standard Deviation); unit: Persons] | 3.62 (1.81) | 3.65 (2.00) | 3.63 (1.91)
Educational Attainment [Count of Participants; unit: Participants]
  Some High School | 3 | 5 | 8
  High School Graduate | 26 | 19 | 45
  Some college/AA degree | 51 | 38 | 89
  Bachelor's Degree | 17 | 31 | 48
  Graduate Degree | 6 | 12 | 18
  Decline to Answer | 1 | 0 | 1
Employment Status (non-exclusive) [Count of Participants; unit: Participants] — Employment Status (non-exclusive). Participants can be counted more than once in the appropriate category.
  Participants
    Student | 37 | 34 | 71
    Full-time work | 42 | 48 | 90
    Part-time work | 26 | 25 | 51
    Full-time homemaker | 3 | 5 | 8
    Unemployed | 10 | 10 | 20
    On leave | 5 | 3 | 8
    Disabled | 3 | 3 | 6
    Other/decline to answer | 3 | 4 | 7
Health Insurance (non-exclusive) [Count of Participants; unit: Participants]
  Private | 53 | 57 | 110
  MediCal/Medicaid | 38 | 43 | 81
  Other public insurance | 13 | 5 | 18
  No Insurance | 2 | 2 | 4
  Don't know | 7 | 2 | 9
  Decline to answer | 1 | 1 | 2
Social Deprivation Index (SDI) [Mean (Standard Deviation); unit: units on a scale] — Social Deprivation Index (SDI) is a composite measure of area level deprivation based on seven demographic characteristics collected in the American Community Survey and used to quantify the socio-economic variation in health outcomes. Total range: 0-100 (Higher values indicate greater social deprivation, representing a worse outcome.)
  units on a scale | 63.11 (27.99) | 63.92 (27.04) | 63.52 (27.46)
Social Vulnerability Index (SVI) [Mean (Standard Deviation); unit: units on a scale] — Social Vulnerability Index (SVI) is a place-based index, database, and mapping application designed to identify and quantify communities experiencing social vulnerability, which refers to the demographic and socioeconomic factors that adversely affect communities that encounter hazards and other community-level stressors. Total range: 0-100 (Higher values indicate greater social vulnerability, representing a worse outcome.)
  units on a scale | 0.57 (0.28) | 0.55 (0.29) | 0.56 (0.29)
Social Needs [Mean (Standard Deviation); unit: units on a scale] — Social Needs is a study-designed questionnaire adapted from the Health Leads Social Needs Screening Tool for assessing various social needs. These needs span categories such as housing, food, transportation, utilities, child care, employment, education, and finances. Total range: 0-10 (higher scores indicate greater social needs).
  citation: Health Leads. (2023). The Health Leads Screening Toolkit. Available at: https://healthleadsusa.org/communications-center/resources/the-health-leads-screening-toolkit/
  units on a scale | 2.13 (1.87) | 2.07 (1.80) | 2.10 (1.83)
T1D diagnosis age [Mean (Standard Deviation); unit: years] | 10.77 (6.01) | 12.22 (5.94) | 11.50 (6.00)
Baseline A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 9.12 (1.44) | 9.26 (1.66) | 9.19 (1.55)
Diabetes device use [Count of Participants; unit: Participants]
  Injections only | 30 | 29 | 59
  Insulin pump only | 12 | 13 | 25
  Injections + CGM | 27 | 20 | 47
  Pump + CGM | 33 | 38 | 71
  Other combination | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6-months in Glycemic Control, Using Glycated Hemoglobin (HbA1C)
Description: HbA1C is a measure of average blood glucose concentration over approximately the previous 12 weeks. HbA1C will be measured using a finger-prick test using the DCA Vantage Analyzer point-of-care system OR AccuBase A1c test with DTI Laboratories. Assessed at Baseline and 6 months; change from baseline to 6 months reported.
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
percentage of glycosylated hemoglobin | -0.44 (1.22) | -0.31 (1.35)

2. Secondary Outcome: Change From Baseline to 6-months Post-test in Diabetes-related Quality of Life, Using the "Audit of Diabetes-Dependent Quality of Life-15" (ADD-QoL-15)
Description: 15-item questionnaire assessing diabetes-related quality of life (qol). Each item contains two parts. Part A is: "If I did not have diabetes, [the question topic] would be", followed by 5 options ranging from "very much better" (or similar; scored as -3) to "worse" (or similar; scored as 1). The fourth option is always "the same" and scored as 0. Part B is: "[the question topic] is" followed by 4 options ranging from "very important" (scored as 3) to "not at all important" (scored as 0). For each question, scores on parts A and B are multiplied, and the 15 products are summed for a total score. Questions 2, 4, 6, 8, 9, & 11 have preliminary yes/no questions, and when a "no" response is given, parts A and B are skipped and the score for that question is 0. The minimum score on each question is -9 and the maximum is 3, with total scores ranging from -135 to 45. Higher/more positive scores represent a better outcome; Lower/ more negative scores represent a worse outcome.
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
score on a scale | 0.39 (1.37) | -0.15 (1.59)

3. Secondary Outcome: Change From Baseline to 6-months Post-test in Diabetes-related Emotional Distress, Using the "Diabetes Distress Scale" (DDS)
Description: 17-item questionnaire assessing diabetes-related emotional distress. Total scores (mean score on all 17 items) range from 1 to 6, with higher scores indicating a worse outcome. Sub-scale scores (emotional burden, physician-related distress, regimen-related distress, and interpersonal distress) each range from 1 to 6, with higher scores indicating a worse outcome. A total or sub-scale score 2.0 - 2.9 should be considered 'moderate distress,' and a total or sub-scale score > 3.0 should be considered 'high distress.'
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
score on a scale | -0.48 (1.01) | -0.25 (1.07)

4. Secondary Outcome: Change in Functional Health and Well-being, Using the "SF-12v2® Health Survey"
Description: Short Form 12-item Health Survey Ver. 2 (SF-12v2) is a 12-item questionnaire assessing functional health & well-being over the last 4 weeks in 8 health domains (physical functioning, role participation with physical health problems, bodily pain, general health, vitality, social functioning, role participation with emotional health problems, mental health), all from the patient's point of view. These 8 domains can be summarized into a physical component summary (PCS) and a mental component summary (MCS). Higher scores indicate a better health state. MCS and PCS scores range from 0-100. Scores are calibrated using general population-derived normative data so that 50 is the avg score or norm. Results can be further summarized into a single preference-based health utility number ranging from 1 (equivalent to perfect health) to 0 (equivalent to being dead), using a complex scoring algorithm (SF-6D) derived from surveying a general U.S. population's preferences for specific health states.
Time Frame: Baseline, 6 months, and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Global Diabetes Self-management, Using the "Diabetes Self-Management Questionnaire-Revised" (DSMQ-R).
Description: 27-item questionnaire assessing self-care activities associated with glycemic control. Higher values indicate more effective self-management. Transformed scores = Actual sum of items / maximum possible sum of items x 10. Total transformed scores range from 0 to 10. Transformed scores on six sub-scales (Dietary control, Glucose management, Glucose monitoring, Medication adherence, Physical activity, and Physician contact) also range from 0 to 10.
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Medication Adherence, Using the "3-item Adherence Self-report Scale" Questionnaire
Description: 3-item questionnaire (Wilson,Lee, Fowler, & Rogers, 2016) assessing adherence to diabetes medication regimen. Item responses for the three adherence items are linearly transformed to a 0-100 scale with zero being the worst adherence, and 100 the best. A total summary score is calculated as the mean of the three individual items, with a range of 0 to 100.
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Self-efficacy for Performing Diabetes Self-management, Using the "Diabetes Empowerment Scale - Short Form" (DES-SF)
Description: 8-item questionnaire assessing self-efficacy for performing diabetes self-management, using 5-point likert scales. The scale is scored by averaging the scores of all completed items. Scores range from 8 to 40, with higher scores indicating higher self-efficacy.
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in Autonomy of Taking Insulin and/or Checking Blood Sugar, Using the "Treatment Self-Regulation Questionnaire" (TSRQ)
Description: 19-item questionnaire, adapted for type 1 diabetes, assessing the degree to which a person's motivation for a particular behavior or a set of behaviors is relatively autonomous or self-determined. Each item can receive a value ranging from 1 - 7 as selected by the participant. The scale has 2 sub-scales: the autonomous regulatory style and the controlled regulatory style. Calculating the scores for the sub-scales consists of averaging the items on that sub-scale. A Relative Autonomous Motivation Index can be formed by subtracting the average for the controlled reasons from the average for the autonomous reasons. Scores range from 1 to 7, with 7 indicating a strong identification with the given autonomy style. The autonomous regulatory style represents the most self-determined form of motivation.
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline to 6-months Post-test in Glycemia, Using Percent Time-in-Range
Description: The percentage of time when blood glucose was between 70 and 180 mg/dl, as measured by a continuous glucose monitor worn for 14 days.
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
percentage of time | 4.44 (22.18) | 1.02 (24.02)

10. Secondary Outcome: Change From Baseline to 6-months Post-test in Glycemia, Using Percent Time in Hyperglycemia
Description: The percentage of time when blood glucose was above 180 mg/dl, as measured by a continuous glucose monitor worn for 14 days.
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
percentage of time | -4.48 (24.68) | -1.61 (26.5)

11. Secondary Outcome: Change From Baseline to 6-months Post-test in Glycemia, Using Percent Time in Hypoglycemia
Description: The percentage of time when blood glucose was below 70 mg/dl, as measured by a continuous glucose monitor worn for 14 days.
Time Frame: Assessed at Baseline and 6 months; change from baseline to 6 months reported
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Lifestyle Intervention | Usual Care
Number analyzed (Participants) | 104 | 105
percentage of time | 0.04 (4.99) | 0.59 (5.09)

12. Secondary Outcome: Change in Cost to Patients
Description: 9 diabetes-related expense questions designed by the study (polar questions, multiple choice, and open-ended). Questions assess loss of income or other productivity due to diabetes (3 items), and impact of cost and health insurance on access to and use of insulin and test strips (6 items).
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in Cost to Payor
Description: 8-item healthcare utilization questionnaire designed by the study. Polar; Yes/No questions about health service usage in the last month: (e.g., "have you had to be admitted to the hospital?"). Open-ended questions about number of time health services were used, (e.g., "how many times were you admitted to the hospital for reasons related to diabetes?").
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months, 10 months, 11 months, and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Description: AE reports reflect a conservative approach to reporting.
Arm/Group | Lifestyle Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 34/104 | 28/105
Other Adverse Events (participants affected / at risk) | 8/104 | 7/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Intervention (N=104) | Usual Care (N=105)
Inpatient Hospitalization: not study related; not hyperglycemia; not hypglycemia (Gastrointestinal disorders) | 2 (2) | 1 (1) — vomiting with blood in it (n=1), or abdominal pain (n=1), or appendicitis (n=1)
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (General disorders) | 0 (0) | 4 (5) — orthostatic hypotension (n=1), or diabetic foot ulcer (n=1), or urinary tract infection + blood clot (n=1), or unknown reason (n=2),
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Infections and infestations) | 0 (0) | 3 (3) — "stomach infection" unrelated to diabetes (n=1), or COVID-19 (n=1), or unknown infection (n=1)
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — ankle fracture
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Psychiatric disorders) | 1 (1) | 1 (1) — mental health issues (further details not known) (n=2)
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Reproductive system and breast disorders) | 0 (0) | 1 (1) — gynecological surgery
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Vascular disorders) | 0 (0) | 1 (1) — stroke
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Gastrointestinal disorders) | 0 (0) | 1 (1) — appendectomy
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Nervous system disorders) | 2 (2) | 0 (0) — seizures (n=1), or MRI for unknown reason (n=1)
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (Cardiac disorders) | 1 (1) | 0 (0) — heart surgery (unrelated to diabetes)
Inpatient Hospitalization: not study related, not hyperglycemia, not hypoglycemia (General disorders) | 1 (1) | 0 (0) — "stress-related diabetes issue"
Severe hypoglycemia (not study-related) -> seizure, loss of consciousness, or emergency transport (Endocrine disorders) | 4 (8) | 7 (10)
Severe hypoglycemia (not study-related) -> seizure, loss of consciousness, or emergency transport (Endocrine disorders) | 1 (1) | 0 (0)
Severe hyperglycemia or diabetic ketoacidosis (not study-related) (Endocrine disorders) | 7 (9) | 8 (13)
Severe hyperglycemia or diabetic ketoacidosis (not study-related) (Endocrine disorders) | 4 (4) | 3 (3)
Severe hyperglycemia or diabetic ketoacidosis (not study-related) (General disorders) | 2 (2) | 2 (2)
Severe hyperglycemia or diabetic ketoacidosis (not study-related) (General disorders) | 2 (2) | 0 (0)
Important medical event based upon appropriate medical judgment (not study-related) (Endocrine disorders) | 0 (0) | 2 (2) — unknown diabetes-related issue (n=1), or loss of consciousness (diabetes-related) (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Gastrointestinal disorders) | 2 (2) | 3 (3) — vomiting due to medication (unrelated to diabetes) (n=1), or "stomach issues" (unrelated to diabetes) (n=1), or appendix or gallbladder issue (unrelated to diabetes) (n=1), or food poisoning/dehydration (n=1), or "gastro" (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (General disorders) | 3 (3) | 10 (10) — swollen foot, retinopathy, chest pain, cocaine overdose/heart problems, diabetic neuropathy, Crohn's disease, car or motorcycle accident, abdominal pain, hand foot and mouth disease, fainting after COVID-19 vaccine, or unknown reason
Important medical event based upon appropriate medical judgment (not study-related) (General disorders) | 3 (3) | 0 (0) — diabetes-related gastroparesis (n=1), or blood clot + urinary tract infection + pancreatitis + gallstones (n=1), or respiratory issues requiring nebulizer (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Immune system disorders) | 0 (0) | 2 (2) — anaphylactic reaction (n=1), or allergic reaction (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Infections and infestations) | 5 (6) | 2 (2) — eye infection (n=1), or kidney infection (unrelated to diabetes) (n=1), or kidney infection (related to diabetes (n=1), or mastitis (n=1), or COVID-19 (n=3), or respiratory syncytial virus (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Infections and infestations) | 3 (3) | 0 (0) — abscess (n=2), or COVID-19 (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) — unknown infection (unrelated to diabetes) (n=1), or food poisoning (n=2)
Important medical event based upon appropriate medical judgment (not study-related) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — food poisoning
Important medical event based upon appropriate medical judgment (not study-related) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — broken patella (n=1), or broken arm (n=1), or broken wrist from horseback riding accident (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — broken arm
Important medical event based upon appropriate medical judgment (not study-related) (Nervous system disorders) | 0 (0) | 1 (1) — concussion (unrelated to diabetes) (n=1)
Important medical event based upon appropriate medical judgment (not study-related) (Surgical and medical procedures) | 0 (0) | 1 (1) — issues with picc line (unrelated to diabetes)
Important medical event based upon appropriate medical judgment (not study-related) (Product Issues) | 1 (1) | 0 (0) — "sensor copper wire lost in stomach" (not from any study-related CGM)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Intervention (N=104) | Usual Care (N=105)
Physical symptom (not serious, not study-related) (Endocrine disorders) | 1 (1) | 0 (0) — low blood sugar levels
Physical symptom (not serious, not study-related) (General disorders) | 0 (0) | 1 (1) — acid reflux, related to diabetes
Physical symptom (not serious, not study-related) (Infections and infestations) | 0 (0) | 2 (2) — stomach flu (n=1), or flu/cold symptoms (n=1)
Physical symptom (not serious, not study-related) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — food poisoning/dehydration
Physical symptom (not serious, not study-related) (Endocrine disorders) | 0 (0) | 1 (1) — hypoglycemia (though no loss of consciousness or seizure)
Physical symptom (not serious, not study-related) (Infections and infestations) | 2 (2) | 0 (0) — cyst/mass (n=1), or walking pneumonia (n=1)
Physical symptom (not serious, not study-related) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — finger injury for shopping cart (n=1), or ankle injury from skateboarding (n=1), or elbow injury/inflammation (n=1)
Physical symptom (not serious, Study-related) (Product Issues) | 1 (1) | 2 (2) — Skin reaction/irritation from study CGM or adhesive tape used to apply study CGM
Psychological symptom (not serious, not study-related) (Psychiatric disorders) | 0 (0) | 1 (1) — stress
Psychological symptom (not serious, Study-related) (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported that they disliked/disagreed with several questions on study questionnaires, especially questions about food because they have an eating disorder.

LIMITATIONS AND CAVEATS:
COVID-19/public health policies may have affected data. COVID-19 led to changes in outcome assessment methods (in-person vs self-administered surveys; Afinion POC vs AccuBase mail-in A1c test) and caused other logistical challenges affecting data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04023487/Prot_SAP_000.pdf